CLINICAL TRIAL: NCT03222674
Title: Multi-center Phase I/II Clinical Trial of Multi-CAR T Cell Therapy for Acute Myeloid Leukemia
Brief Title: Multi-CAR T Cell Therapy for Acute Myeloid Leukemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shenzhen Geno-Immune Medical Institute (Other)
Collaborators: Zhujiang Hospital, Southern Medical University, Guangzhou, Guangdong, China (Unknown); Yunnan Cancer Hospital (Other)
Responsible Party: Principal Investigator, Lung-Ji Chang, President, Shenzhen Geno-Immune Medical Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: GIMI-IRB-17015
Record Dates: First submitted 2017-07-14; First posted 2017-07-19 (Actual); Last update posted 2018-10-17 (Actual); Status verified 2018-10

CONDITIONS: Acute Myeloid Leukemia
Keywords: AML; CAR T; Muc1,CLL1, CD33, CD38, CD56, and/or CD123
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Single arm (Experimental): CAR T cells to treat AML
  Interventions: Biological: Muc1/CLL1/CD33/CD38/CD56/CD123-specific gene-engineered T cells

INTERVENTIONS:
Biological: Muc1/CLL1/CD33/CD38/CD56/CD123-specific gene-engineered T cells — Infusion of Muc1/CLL1/CD33/CD38/CD56/CD123-specific gene-engineered T cells

SUMMARY:
The purpose of this clinical trial is to assess the feasibility, safety and efficacy of multi-CAR T cell therapy targeting different AML surface antigens in patients with relapsed or refractory acute myeloid leukemia (AML). Another goal of the study is to learn more about the function of the multi-CAR T cells and their persistency in the patients.

DETAILED DESCRIPTION:
Acute myeloid leukemia (AML) is a malignant disease characterized by the rapid growth of myeloblasts that build up in the bone marrow and interfere with the production of normal blood cells.

In this study, the patients' own T cells will be genetically modified with lentiviral vectors expressing chimeric antigen receptors. The multi-CAR T cells recognize specific molecules such as CD33, CD38, CD123, CD56, MucI, and CLL1, which are often found expressed on the surface of AML cells. The engineered CAR T cells will be infused into patients.

The purpose of this clinical study is to assess the feasibility, safety and efficacy of the multi-CAR T cell therapy against AML. Another goal of the study is to learn more about the function of the multi-CAR T cells and their persistency in the patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age older than 2 years.
2. CD33, CD38, CD56, CD123, MucI, and CLL1 expression can be identified in the malignant cells by immuno-histochemical staining or flow cytometry.
3. Karnofsky performance status (KPS) score is higher than 80 and life expectancy > 2 months.
4. Adequate bone marrow, liver and renal function as assessed by the following laboratory requirements: cardiac ejection fraction ≥ 50%, oxygen saturation ≥ 90%, creatinine ≤ 2.5 × upper limit of normal, aspartate aminotransferase (AST) and alanine aminotransferase (ALT) ≤ 3 × upper limit of normal, total bilirubin ≤ 2.0mg/dL.
5. Hgb≥80g/L.
6. No cell separation contraindications.
7. Abilities to understand and the willingness to provide written informed consent.

Exclusion Criteria:

1. Sever illness or medical condition, which would not permit the patient to be managed according to the protocol, including active uncontrolled infection.
2. Active bacterial, fungal or viral infection not controlled by adequate treatment.
3. Known HIV or hepatitis B virus (HBV) infection.
4. Pregnant or nursing women may not participate.
5. History of glucocorticoid for systemic therapy within the week prior to entering the test.
6. Previously treatment with any gene therapy products.
7. Patients, in the opinion of investigators, may not be eligible or not able to comply with the study.

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 10 (Estimated)
Dates: Start 2017-07-15 (Actual); Primary Completion 2019-12-31 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
percentage of patients with treatment related adverse effect | a year
  percentage of participants with treatment-related adverse events, as assessed by physical exam, vital signs, standard clinical labs and so on.

SECONDARY OUTCOMES:
Anti tumor activity of fourth generation CAR-T cells in patients with relapsed or refractory AML | a year
  scale of CAR copies and leukemic cell burden (for efficacy)

CONTACTS AND LOCATIONS:
Overall Officials: Lung-Ji Chang, Principal Investigator — Shenzhen Geno-Immune Medical Institute
Locations (3):
- China (3):
  - Zhujiang Hospital of Southern Medical University, Guangzhou, Guangdong
  - Shenzhen Geno-immune Medical Institute, Shenzhen, Guangdong
  - Yunnan Cancer Hospital & The Third Affiliated Hospital of Kunming Medical University & Yunnan Cancer Center, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Pei K, Xu H, Wang P, Gan W, Hu Z, Su X, Zhang H, He Y. Anti-CLL1-based CAR T-cells with 4-1-BB or CD28/CD27 stimulatory domains in treating childhood refractory/relapsed acute myeloid leukemia. Cancer Med. 2023 Apr;12(8):9655-9661. doi: 10.1002/cam4.5916. Epub 2023 Apr 9. PMID 37031462